CLINICAL TRIAL: NCT00397787
Title: A Phase II Study of Sunitinib Malate (SU11248, NSC #736511, IND #74,019) in Patients With Previously Treated Pancreatic Adenocarcinoma With Measurable Metastatic Disease Following Progression on Front-Line Gemcitabine-Based Therapy
Brief Title: Sunitinib in Treating Patients With Metastatic Pancreatic Cancer That Progressed After First-Line Therapy With Gemcitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02823; CALGB-80603; U10CA031946 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sunitinib

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive oral sunitinib malate daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with metastatic pancreatic cancer that progressed after first-line therapy with gemcitabine. Sunitinib may stop the growth of pancreatic cancer by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate to sunitinib malate in patients with previously treated metastatic pancreatic adenocarcinoma.

SECONDARY OBJECTIVES:

I. To determine the duration of response, progression-free survival and overall survival of sunitinib malate in patients with previously treated metastatic pancreatic adenocarcinoma.

II. To determine the safety of sunitinib malate in patients with previously treated metastatic pancreatic adenocarcinoma.

OUTLINE: This is a multicenter, nonrandomized study.

Patients receive oral sunitinib malate daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed every 3 months until 2 years from study entry or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic documentation of pancreatic adenocarcinoma with evidence of disease progression following first-line therapy is required
* No brain metastases
* Patients with measurable disease

  * Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded as >= 20 mm with conventional techniques or as>= 10 mm with spiral computed tomography (CT) scan; of particular note, the primary pancreatic tumor does not constitute measurable disease; therefore, patients with locally advanced pancreatic cancer as the sole site of disease are not eligible
* Patients must have received one of the following prior therapies containing gemcitabine:

  * One and only one prior therapy for metastatic disease with gemcitabine, or a gemcitabine-containing cytotoxic combination, or
  * One prior chemoradiation therapy containing gemcitabine for inoperable locally advanced pancreatic cancer, as long as the patient has subsequently progressed and has measurable disease outside a radiation port, or
  * One prior adjuvant chemotherapy regimen or chemoradiation therapy containing gemcitabine if the patient subsequently progressed within 3 months of completion of adjuvant therapy; patients who have received chemoradiation in the adjuvant setting must have measurable disease outside the radiation port
* No prior therapy with any other antiangiogenic agent (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, PTK787, VEGF Trap, etc.)
* At least 4 weeks must have elapsed prior to initiation of treatment since the completion of chemotherapy and/or radiation therapy
* At least 4 weeks must have elapsed prior to registration since any major surgery
* Prior erlotinib is permitted; the last dose must have been administered 14 or more days prior to initiation of treatment; all erlotinib related side effects must have resolved to < grade 1 prior to registration
* No significant cardiac disease including:

  * QTc prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant EKG abnormalities
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to registration
  * History of class III or IV heart failure within 12 months prior to registration as defined by the NYHA functional classification system
* In addition, patients with history of hypertension must be well controlled (< 140/90) on a regimen of anti-hypertensive therapy
* Patients with a history of hypothyroidism are eligible, provided they are currently euthyroid
* The use of inhibitors and inducers of CYP3A4 is not permitted:

  * The following inhibitors of CYP3A4 is prohibited within 7 days before beginning and during treatment with sunitinib:

    * Azole antifungals (ketoconazole, itraconazole)
    * Diltiazem
    * Clarithromycin
    * Erythromycin
    * Verapamil
    * Delavirdine
    * HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir)
  * The following inducers of CYP3A4 are prohibited within 12 days before beginning and during treatment with sunitinib:

    * Rifampin
    * Rifabutin
    * Carbamazepine
    * Phenobarbital
    * Phenytoin
    * St. John's wort
    * Efavirenz
    * Tipranavir
  * Other inhibitors or inducers of CYP3A4 may be used if necessary, but their use is discouraged
* The use of agents with proarrhythmic potential (e.g., quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, flecainide) is not permitted during the study
* ECOG performance status 0-2
* No history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to registration
* No history of pulmonary embolism within the past 6 months
* Patients who require use of therapeutic doses of coumadin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; Note: Low molecular weight heparin is permitted provided the patient's PT INR is < 1.5
* No serious or non-healing wound, ulcer, or bone fracture
* No history (within 6 months) of significant bleeding events (e.g., upper or lower GI bleeding, hemoptysis, or hematuria), abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
* No evidence of duodenal invasion by the tumor on CT scan
* No "currently active" second malignancy other than non-melanoma skin cancers; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse
* Non-pregnant and not breast feeding; pregnant women are excluded from this study because sunitinib is an antiangiogenic agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib, breastfeeding should be discontinued if the mother is treated with sunitinib malate
* ANC >= 1,500/μl
* Platelet count >= 100,000/μl
* Bilirubin < 1.5 mg/dL
* PT and PTT =< 1.5 X ULN
* Creatinine =< 1.5 mg/dL
* AST (SGOT) =< 2.5 X ULN if no liver metastases (=< 5 X ULN if liver metastases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Response (CR/PR/stable disease) as measured by RECIST criteria | At 6 weeks post-initiation of protocol treatment

SECONDARY OUTCOMES:
Response duration | Up to 2 years
  Duration of response will be determined for the subset of patients who achieve a confirmed response of CR or PR. Duration of objective response will be defined as the time from the first tumor assessment indicating response (later confirmed) to the time of disease progression or death from any cause.
Progression-free survival (PFS) | Up to 2 years
  Median and 1-year survival will be assessed using Kaplan-Meier methods.
Number and percentage of patients reporting common and serious adverse events (AEs), the AEs related to sunitinib, reason for study discontinuation, clinically significant laboratory abnormalities, and AEs with worst NCI CTCAE grade | Up to 2 years
  Summarized descriptively for all patients receiving at least one dose of sunitinib.
Overall survival (OS) | Up to 2 years
  Median and 1-year survival will be assessed using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Cancer and Leukemia Group B, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] O'Reilly EM, Niedzwiecki D, Hall M, Hollis D, Bekaii-Saab T, Pluard T, Douglas K, Abou-Alfa GK, Kindler HL, Schilsky RL, Goldberg RM; Cancer and Leukemia Group B. A Cancer and Leukemia Group B phase II study of sunitinib malate in patients with previously treated metastatic pancreatic adenocarcinoma (CALGB 80603). Oncologist. 2010;15(12):1310-9. doi: 10.1634/theoncologist.2010-0152. Epub 2010 Dec 10. PMID 21148613